CLINICAL TRIAL: NCT02920463
Title: DetermInants of Antimicrobial Use aNd De-escalAtion in Critical Care (DIANA Study)
Brief Title: DetermInants of Antimicrobial Use aNd De-escalAtion in Critical Care (DIANA)
Acronym: DIANA
Status: Completed | Type: Observational
Sponsor: University Hospital, Ghent (Other)
Responsible Party: Sponsor
Other Study IDs: EC/2016/0938
Record Dates: First submitted 2016-08-26; First posted 2016-09-30 (Estimated); Last update posted 2019-09-20 (Actual); Status verified 2019-09

CONDITIONS: Infection
Keywords: Anti-Infective agents; Antimicrobial stewardship; Empirical antibiotic therapy; De-escalation; Critical care
MeSH Terms: conditions — Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Critically ill patients with infection: Critically ill adult patients receiving empirical antibiotic therapy for suspected or confirmed infections at the Intensive Care Unit

SUMMARY:
DetermInants of Antimicrobial use aNd de-escalAtion in critical care (DIANA study), is a multicenter, international, prospective, observational cohort study, aiming to describe the rate of de-escalation as well as the associated outcome and the empirical antibiotic therapy for infections at the intensive care unit.

DETAILED DESCRIPTION:
Despite the consensus regarding spectrum and timing of antibiotic therapy, antimicrobial use varies across ICUs; indeed there are important variations in choice, dosing, method of administration, duration of antimicrobial therapy and de-escalation of empirical therapy. DetermInants of Antimicrobial use aNd de-escalAtion in critical care (DIANA study), is a multicenter, international, prospective, observational cohort study, aiming to describe the rate of de-escalation as well as the associated outcome and the empirical antibiotic therapy for infections at the intensive care unit.

Given the explorative nature of this study the required number of patients was not calculated. The investigators aim to include 2000 patients in whom empirical antibiotics are started. With an estimated de-escalation rate of 35%, an estimation to include 700 patients in whom de-escalation is performed is made which would allow for a suitable multivariable analysis.

For each participating center center data will be collected as detailed in an electronic Center Report Form. This will be completed only once per center.

For each participating center data on 4 elements will be collected: ICU-related data, microbiology laboratory practices, definition of de-escalation as used in the participating center and local de-escalation practices, background resistance levels.

This is a prospective observational study in which patients will be included in the participating centers during a 2-week period.

For each patient included in the study, data will be collected in an electronic Case Report Form.

For each included patient data on 4 elements will be collected: patient data (demographics, underlying and co-morbid conditions, patient characteristics on different time points), infection data (clinical and microbiological), treatment data (antimicrobial therapy and source control) and outcome data (28 day follow up period)

National coordinators:

National Coordinators will be appointed by the Steering Committee and will have a key role in the conduction of the study in the individual countries as leaders of the project.

Ethics committee approval:

Ethics committee approval may vary from country to country. The national coordinator is responsible for obtaining ethics committee approval if this is required on a national level (or any procedure similar to this). Informed consent will be obtained from the subject or nominated representative (where applicable). As this is an observational study some countries and sites may waive the need for informed consent.

Data management:

All patient data will be collected anonymously and will be entered in an electronic data capturing system. Data provided by the local investigators are primarily the property of the ICU that collected the data. Local investigators shall have access to their data after they have been entered in the central database.The servers of the system are hosted at True; True has been certified by the Lloyd's Register Quality Assurance (LRQA) according to the international information security norm ISO 27001:2013. True provides its services in accordance with the NEN7510 norm for information security in healthcare.

Data control:

Local investigators may be contacted for queries in case of outliers, excessive missing values and other reasons deemed relevant by the primary investigator.

Statistical analysis:

Statistical analysis will be performed by the primary investigators using a statistical software program and assisted by expert statisticians when necessary.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older.
* Patient is admitted to an ICU and has an anticipated need of ICU support of at least 48 hours.
* Patient has a suspected or confirmed bacterial infection (community-, healthcare-, hospital- or ICU-acquired).
* Empirical antibiotic therapy is started for this infection at any time in the ICU or no more than 24 hours prior to ICU admission. If the initial antibiotic therapy is considered inadequate and another empirical scheme is chosen at ICU admission, this will be the empirical antibiotic of the study.
* Causative pathogen and susceptibility are unidentified at time of initiation of the antibiotic therapy (Gram staining results may be known).
* Signed informed consent (if required by local ethics committee).

Exclusion Criteria:

* Previous inclusion in this study for another infection - each patient can only be included once.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients admitted to the intensive care unit during a 2-week period between October 2016 and December 2017. Participating centers can select the weeks of participation based on local considerations and staff availability.All consecutive patients that are eligible according to inclusion and exclusion criteria should be included in the study.
Sampling Method: Probability Sample
Enrollment: 1495 (Actual)
Dates: Start 2016-10-01 (Actual); Primary Completion 2018-06-30 (Actual); Study Completion 2018-06-30 (Actual)

PRIMARY OUTCOMES:
Number of patients in which the empirical antibiotic therapy is de-escalated | 28 days
  Included patients will be monitored for 28 days. This is the number of patients in which the empirical antibiotic therapy is de-escalated during the time of observation.
Proportion of patients with clinical cure at day 7 in de-escalated patients versus non-deescalated patients | 7 days
  This is the proportion of patients in which the infection under study is clinically cured, which is defined as: 'disappearance of all signs and symptoms related to the infection under study' in de-escalated versus non-deescalated patients.

SECONDARY OUTCOMES:
Antibiotics used in empirical antimicrobial therapy in critically ill patients | 28 days
  Which antibiotic categories are chosen empirically to treat the infection under study in all critically ill patients included during the study period.
Proportion of appropriate empirical antibiotic therapy in critically ill patients | 28 days
  This is the proportion of all empirical antibiotic prescriptions that has in-vitro activity against all causative pathogens.
Antibiotics used in definitive antimicrobial therapy in critically ill patients | 28 days
  Which antibiotic categories are chosen as definitive antimicrobial therapy to treat the infection under study in all critically ill patients included during the study period.
Duration of antimicrobial treatment for the infection under study in de-escalated patients versus non-deescalated patients | 28 days
Duration of hospitalization on the intensive care unit in de-escalated patients versus non-deescalated patients | 28 days
Number of antibiotic free days in de-escalated patients versus non-deescalated patients | 28 days
Proportion of patients who died at day 28 in de-escalated patients versus non-deescalated patients | 28 days
Proportion of patients in whom drug-resistant pathogens emerge in de-escalated patients versus non-deescalated patients | 28 days
  Included patients will be monitored for 28 days. This is the proportion of multidrug resistant, extensively drug-resistant, pandrug- resistant pathogens and pathogens resistant to the administered empirical antibiotic therapy that emerge in de-escalated patients versus non-deescalated patients
Proportion of patients with infection relapse, superinfections and subsequent infections in de-escalated patients versus non-deescalated patients | 28 days
  Infection relapse being defined as an infection occurring after stopping all antimicrobial agents for the primary infection under study with the same causative microorganism (a different susceptibility pattern may be present).
  Subsequent infection being defined as an infection occurring after stopping all antimicrobial agents for the primary infection under study, with a different causative microorganism.
  Superinfection being defined as an infection superimposed on the primary infection under study with a different causative microorganism.
Proportion of antimicrobial prescriptions in which a loading dose is used | 28 days
Proportion of antimicrobial prescriptions which are administered in a continuous or extended infusion | 28 days

CONTACTS AND LOCATIONS:
Overall Officials: Jan J De Waele, MD,PhD, Principal Investigator — University Hospital, Ghent
Locations (1):
- Ghent University Hospital, Ghent, Belgium

IPD SHARING:
Plan to Share IPD: Yes
Data will be shared with participating centers only. Data provided by the local investigators are primarily the property of the ICU that collected the data. Local investigators shall have access to their data after they have been entered in the central database.

REFERENCES:
- [Background] Tabah A, Cotta MO, Garnacho-Montero J, Schouten J, Roberts JA, Lipman J, Tacey M, Timsit JF, Leone M, Zahar JR, De Waele JJ. A Systematic Review of the Definitions, Determinants, and Clinical Outcomes of Antimicrobial De-escalation in the Intensive Care Unit. Clin Infect Dis. 2016 Apr 15;62(8):1009-1017. doi: 10.1093/cid/civ1199. Epub 2015 Dec 23. PMID 26703860
- [Background] Leone M, Bechis C, Baumstarck K, Lefrant JY, Albanese J, Jaber S, Lepape A, Constantin JM, Papazian L, Bruder N, Allaouchiche B, Bezulier K, Antonini F, Textoris J, Martin C; AZUREA Network Investigators. De-escalation versus continuation of empirical antimicrobial treatment in severe sepsis: a multicenter non-blinded randomized noninferiority trial. Intensive Care Med. 2014 Oct;40(10):1399-408. doi: 10.1007/s00134-014-3411-8. Epub 2014 Aug 5. PMID 25091790
- [Derived] Yoshida H, Motohashi T, De Bus L, De Waele J, Takaba A, Kuriyama A, Kobayashi A, Tanaka C, Hashi H, Hashimoto H, Nashiki H, Shibata M, Kanamoto M, Inoue M, Hashimoto S, Katayama S, Fujiwara S, Kameda S, Shindo S, Suzuki T, Komuro T, Kawagishi T, Kawano Y, Fujita Y, Kida Y, Hara Y, Fujitani S; DIANA Study Japanese group. Use of broad-spectrum antimicrobials for more than 72 h and the detection of multidrug-resistant bacteria in Japanese intensive care units: a multicenter retrospective cohort study. Antimicrob Resist Infect Control. 2022 Sep 29;11(1):119. doi: 10.1186/s13756-022-01146-3. PMID 36175948
- See also: Click here for more information about this study: DetermInants of Antimicrobial use aNd de-escalAtion in critical care — http://www.dianastudy.ugent.be